CLINICAL TRIAL: NCT04006054
Title: Cerebral Protection of Dexmedetomidine Against Paroxysmal Sympathetic Overexcited in Patients With Traumatic Brain Injury
Brief Title: Study on Cerebral Protection of Dexmedetomidine for Patients With Traumatic Brain Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019040111
Record Dates: First submitted 2019-06-13; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine treatment group (Experimental): Dexmedetomidine will be administrated at a dose of 0.25-0.75 µg/(kg*h) for 5 days
  Interventions: Drug: Dexmedetomidine
- Midazolam treatment group (Active Comparator): Midazolam will be administrated at a dose of 0.25-0.75 µg/(kg*h) for 5 days
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — When the patients who suffered traumatic brain injury are in NICU，Dexmedetomidine is given for sedation about 5 days .
  Other Names: DG
  Arms: Dexmedetomidine treatment group
Drug: Midazolam — When the patients who suffered traumatic brain injury are in NICU，Midazolam is given for sedation about 5 days .
  Other Names: MG
  Arms: Midazolam treatment group

SUMMARY:
The aim of the study is to investigate whether dexmedetomidine could suppress catecholamine release into peripheral blood to prevent PSH attacks and to achieve neuroprotection.

DETAILED DESCRIPTION:
Paroxysmal sympathetic hyperactivity (PSH) is a syndrome typically recognized in patients suffering from traumatic brain injury, characterized by paroxysmal increases in sympathetic activity such as elevated heart rate, increased blood pressure and respiratory rate, high temperature, excessive sweating and abnormal motor (posturing) activity.

This prospective study will include patients with traumatic brain injury,who will be divided into two groups, evaluated by the Paroxysmal Sympathetic Hyperactivity-Assessment Measure (PSH-AM). Patients will also be evaluated with head CT.

The aim of the study is to investigate whether dexmedetomidine could suppress catecholamine release into peripheral blood to prevent PSH attacks and to achieve neuroprotection.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years
2. Moderate or severe traumatic brain injury
3. GCS≤12
4. Diagnosed by CT
5. No catecholamines (such as dopamine, adrenaline, norepinephrine) have been used before admission
6. Have a clear history of head trauma
7. Non-open traumatic brain injury

Exclusion Criteria:

1. Severe liver dysfunction (Child-Pugh B or C)
2. Severe renal dysfunction (serum creatinine > 445 mmol / L or blood urea nitrogen > 20 mmol / L)
3. Hemodynamic instability when entering the ICU (heart rate <50 beats / min or hypotension, SBP <90mmHg or MAP <65mmHg)
4. Deaths within 72 hours after entering the ICU
5. Severe multiple injuries (ISS≥25 points)
6. Have central nervous system diseases (such as hypoxic ischemic encephalopathy, stroke, brain tumors, etc.)
7. Allergic to dexmedetomidine or midazolam
8. Observed with the results of disease interference test (such as pheochromocytoma, etc.)
9. In pregnancy or lactation
10. Receiving hypothermia treatment
11. Are participating in other drug research or clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Epinephrine | At admission (baseline)
  Epinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Epinephrine | 24 hours after injury
  Epinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Epinephrine | 48 hours after injury
  Epinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Epinephrine | 72 hours after injury
  Epinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Norepinephrine | At admission (baseline)
  Norepinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Norepinephrine | 24 hours after injury
  Norepinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Norepinephrine | 48 hours after injury
  Norepinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.
Norepinephrine | 72 hours after injury
  Norepinephrine is a hormone secreted by the body.When the patient suffers brain injury, the concentration of Epinephrine will increase significantly.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No